CLINICAL TRIAL: NCT04785521
Title: Glutamate Excitotoxicity in Brain Metastases From Lung, Breast and Melanoma Treated With Stereotactic Radiosurgery
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Pietro Mortini, MD, Prof., Head of department, IRCCS San Raffaele
Other Study IDs: NCH04-2020
Record Dates: First submitted 2021-03-02; First posted 2021-03-08 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Brain Metastases, Adult
Keywords: Brain metastases; Glutamate; Stereotactic radiosurgery
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- BM patients: Adult patients carrying new diagnosed BM confirmed by MRI
  Interventions: Radiation: Stereotactic radiosurgery; Diagnostic Test: Blood samples
- No BM patients: Adult patients carrying extracranial tumor without BM as confirmed by MRI
  Interventions: Diagnostic Test: Blood samples
- Benign lesion patients: Adult patients carrying intracranial extra-axial tumor as as confirmed by MRI
  Interventions: Radiation: Stereotactic radiosurgery; Diagnostic Test: Blood samples

INTERVENTIONS:
Radiation: Stereotactic radiosurgery — Gamma Knife stereotactic radiosurgery (SRS-GK)
  Groups: BM patients; Benign lesion patients
Diagnostic Test: Blood samples — Serum Glu levels and Glu-regulation markers assessed prior to and following SRS-GK in BM or benign lesions or at baseline in non-BM patients.

SUMMARY:
Brain metastases (BM) represents a devastating clinical reality, carrying an estimated survival time of less than one year. Number of reasons, including complicated tumor biology and difficulties in modeling metastatic cancer in brain microenvironment, do hinder research on this topic. BM are indeed the most frequent neoplasm in the central nervous system (CNS) and is estimated that up to 14% of all newly diagnosed cancers will metastasize to the brain. A number of reasons, including complicated tumor biology and difficulties in modeling metastatic cancer in brain microenvironment, do hinder research on this topic. Present knowledge regarding alterations in Glutamate (Glu) homeostasis and BM is poor. This study aims at investigating Glu balance in BM patients and providing supporting evidence to the identification of new putative biomarkers to be used as potential therapeutic targets.

DETAILED DESCRIPTION:
Experimental procedure:

Serum levels of glutamic oxaloacetic transaminase (GOT1), glutamate Pyruvate Transaminase (GPT) and lactate dehydrogenase (LDH) levels and serum glutamate, aspartate and lactate levels of a total of 100 patients will be collected and divided in three different groups:

* A: BM group (n=50), patients affected by BM from lung, breast and melanoma, candidates to SRS
* B: Control group 1 (n=25), patients with the same primary controlled tumors without nor brain nor extracranial metastases
* C: Control group 2 (n=25), patients with benign intracranial lesions candidates to SRS treatment.

In A) and C) serum GOT1, GPT and LDH levels and serum glutamate, aspartate, lactate levels will be evaluated before and after SRS treatment (at 3, 6 and 9 months follow-up).

In B) serum biomarkers levels will be only collected at baseline.

• Oncological and imaging data will be collected during follow-up in patients enrolled in the present studies. MRI imaging will be performed at definite timepoints (baseline and 3, 6 and 9 months follow-up).

Serum levels of markers will be analyzed in each group and results will be compared between them. Moreover, MRI changes and oncological relevant outcomes will be investigated.

ELIGIBILITY:
Inclusion Criteria (Target group)

* Adult patients carrying melanoma, breast or lung cancer BM of new diagnosis
* Patients eligible to SRS-GK treatment

Inclusion Criteria (Control group 1)

- Adult patients carrying melanoma, breast or lung cancer without BM

Inclusion Criteria (Control group 2)

* Adult patients carrying intracranial extra-axial benign tumor
* Patients eligible to SRS-GK treatment

Exclusion Criteria:

* Acute or chronic liver disease
* Severe anemia (Hb <8g/dl)
* Pregnant or breastfeeding patient
* Pediatric patients
* Patients not able to express informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Target group:
  Adult patients affected by melanoma, breast or lung cancer BM of new diagnosis as confirmed by MRI ongoing SRS-GK treatment.
  Control group 1:
  Adult patients affected by melanoma, breast or lung cancer without BM.
  Control group 2:
  Adult patients affected by intracranial extra-axial benign tumor as confirmed by MRI ongoing SRS-GK treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum markers determination in newly diagnosed BM (lung, breast and melanoma) patients, before SRS treatment. | Baseline (pre-SRS);
  GOT1, GPT and LDH levels and serum glutamate, aspartate and lactate levels. All measures in mg/dl.
Serum markers determination in newly diagnosed BM (lung, breast and melanoma) patients, after SRS treatment. | Baseline (pre-SRS) and at 3, 6 and 9 months
  GOT1, GPT and LDH levels and serum glutamate, aspartate and lactate levels. All measures in mg/dl.
Serum markers determination in melanoma, lung or breast cancer patients without BM. | Baseline
  Comparison of serum GOT1, GPT and LDH levels and serum glutamate, aspartate and lactate levels between BM and non-BM patients. All measures in mg/dl.
Serum markers determination in patients carrying benign intracranial lesions before and after SRS treatment. | Baseline (pre-SRS) and at 3, 6 and 9 months
  Comparison of serum GOT1, GPT and LDH levels and serum glutamate, aspartate and lactate levels between BM and benign lesion patients. All measures in mg/dl.

SECONDARY OUTCOMES:
Studying correlation of serum markers levels with MRI changes following SRS-GK | 3, 6 and 9 months
  Correlation between trends of markers and incidence of MRI changes.

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Mortini, MD, Prof., Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lowery FJ, Yu D. Brain metastasis: Unique challenges and open opportunities. Biochim Biophys Acta Rev Cancer. 2017 Jan;1867(1):49-57. doi: 10.1016/j.bbcan.2016.12.001. Epub 2016 Dec 6. PMID 27939792
- [Background] Franzin A, Snider S, Picozzi P, Bolognesi A, Serra C, Vimercati A, Passarin O, Mortini P. Evaluation of different score index for predicting prognosis in gamma knife radiosurgical treatment for brain metastasis. Int J Radiat Oncol Biol Phys. 2009 Jul 1;74(3):707-13. doi: 10.1016/j.ijrobp.2008.08.062. Epub 2008 Dec 25. PMID 19095375
- [Background] Robert SM, Sontheimer H. Glutamate transporters in the biology of malignant gliomas. Cell Mol Life Sci. 2014 May;71(10):1839-54. doi: 10.1007/s00018-013-1521-z. Epub 2013 Nov 27. PMID 24281762
- [Background] Miladinovic T, Nashed MG, Singh G. Overview of Glutamatergic Dysregulation in Central Pathologies. Biomolecules. 2015 Nov 11;5(4):3112-41. doi: 10.3390/biom5043112. PMID 26569330
- [Background] Sharma MK, Seidlitz EP, Singh G. Cancer cells release glutamate via the cystine/glutamate antiporter. Biochem Biophys Res Commun. 2010 Jan 1;391(1):91-5. doi: 10.1016/j.bbrc.2009.10.168. Epub 2009 Nov 5. PMID 19896463
- [Background] Zeng Q, Michael IP, Zhang P, Saghafinia S, Knott G, Jiao W, McCabe BD, Galvan JA, Robinson HPC, Zlobec I, Ciriello G, Hanahan D. Synaptic proximity enables NMDAR signalling to promote brain metastasis. Nature. 2019 Sep;573(7775):526-531. doi: 10.1038/s41586-019-1576-6. Epub 2019 Sep 18. PMID 31534217
- [Background] Willard SS, Koochekpour S. Glutamate signaling in benign and malignant disorders: current status, future perspectives, and therapeutic implications. Int J Biol Sci. 2013 Aug 9;9(7):728-42. doi: 10.7150/ijbs.6475. eCollection 2013. PMID 23983606